CLINICAL TRIAL: NCT03492177
Title: A Prospective, Multicenter, Open Label, Single Arm, Phase 2 Study to Investigate the Safety, Tolerability and Pharmacokinetics of Selexipag in Children With Pulmonary Arterial Hypertension
Brief Title: A Clinical Study of to Confirm the Doses of Selexipag in Children With Pulmonary Arterial Hypertension
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-065A203; AC-065A203 (Other: Janssen Research & Development, LLC); 2022-503042-42-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pediatric
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- open label selexipag (Experimental): The first dose of selexipag (Uptravi) will be administered in the evening of Day 1 and will be based on the body weight. Thereafter selexipag will be administered twice daily (morning and evening). Selexipag will be up-titrated during the first 12 weeks, with weekly increments equal to the starting dose until the participants reach their individual maximum tolerated dose (iMTD) or until a maximum dose corresponding to their baseline weight category is achieved (which will be 8-fold of the corresponding starting dose). Up-titration is followed by a stable maintenance treatment period from Week 12 to Week 16, at the maximum tolerated dose. Thereafter, participants will be treated with selexipag as long as the treatment is beneficial to the participants, as per investigator's decision.
  Interventions: Drug: selexipag (Uptravi)

INTERVENTIONS:
Drug: selexipag (Uptravi) — Film-coated tablets for oral administration
  Other Names: ACT-293987; JNJ-67896049

SUMMARY:
The purpose of this study to confirm the selexipag starting dose(s), selected based on pharmacokinetic (PK) extrapolation from adults, that leads to similar exposure as adults doses in children from greater than or equal to (>=) 2 to less than (˂) 18 years of age with Pulmonary Arterial Hypertension (PAH), by investigating the PK of selexipag and its active metabolite ACT-333679 in this population.

DETAILED DESCRIPTION:
The selection of the starting dose for pediatric participants is based on the PK extrapolation from adults, taking into account the children body weight category, in order to lead to an exposure similar to that in adult PAH participants at a starting dose of 200 micrograms (mcg). As in adults, selexipag will be up-titrated to the individual maximum tolerated dose (iMTD) during the first 12 weeks. Approximately 60 participants will be enrolled in 3 different age cohorts to obtain at least 45 participants with evaluable PK profiles: Cohort 1: >= 12 to < 18 years of age, Cohort 2: >= 6 to < 12 years of age, Cohort 3: >= 2 to < 6 years of age. In each age cohort the starting dose will depend on the body weight. Enrollment will start with both Cohort 1 and Cohort 2. After completion of PK assessments in at least 15 participants from Cohort 1 at Week 12, a first interim analysis will be conducted to establish the dose-exposure relationship using a population PK model. The PK data from any participants in Cohort 2 who have completed their PK assessments at this time will be included in this first interim analysis. Results of this model-based analysis will be used to confirm or adjust the selexipag doses initially selected. Enrollment of Cohort 3 (children >= 2 to < 6 years of age) will start once the appropriate doses have been confirmed in a second interim analysis of PK data from Cohorts 1 and 2, and if there is no safety concern based on review by an Independent Data Monitoring Committee (IDMC).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent by the parent(s) or Legally authorized representative(s) AND assent from developmentally capable children
* Males or females between greater than or equal to (>=) 2 and less than (<) 18 years of age with weight >= 9 kilograms (kg)
* Pulmonary arterial hypertension (PAH) diagnosis confirmed by documented historical right heart catheterization (RHC) performed at any time before participant's enrollment
* PAH with one of the following etiologies:

  * idiopathic (iPAH),
  * heritable (hPAH),
  * associated with congenital heart disease (CHD): PAH with co-incidental CHD; post-operative PAH (persisting/ recurring/ developing >= 6 months after repair of CHD)
  * Drug or toxin-induced
  * PAH associated with HIV
  * PAH associated with connective tissue disease
* Word Health Organization functional class (WHO FC) II to III
* Participants treated with an endothelin receptor antagonist (ERA) and/or a phosphodiesterase type 5 (PDE-5) inhibitor provided that the treatment dose(s) has been stable for at least 3 months prior to enrollment, or participants who are not candidates for these therapies
* Females of childbearing potential must have a negative pregnancy test at Screening and at Enrollment, and must agree to undertake monthly pregnancy tests, and to use a reliable method of contraception (if sexually active) from screening up to study drug discontinuation plus 30 days (EOS)

Key Exclusion Criteria:

* Participants with PAH due to portal hypertension, schistosomiasis, pulmonary veno-occlusive disease (PVOD) and/or pulmonary capillary hemangiomatosis
* Participants with PAH associated with Eisenmenger syndrome
* Participants with moderate to large left-to-right shunts
* Participants with cyanotic congenital cardiac lesions such as transposition of the great arteries, truncus arteriosus, univentricular heart or pulmonary atresia with ventricular septal defect, as well as Participants with Fontan-palliation
* Participants with pulmonary hypertension due to lung disease
* Previous treatment with Uptravi (selexipag) within 2 weeks prior to enrollment
* Participants having received prostacyclin (epoprostenol) or prostacyclin analogs (that is, treprostinil, iloprost, beraprost) within 2 months prior to enrollment or are scheduled to receive any of these compounds during the trial
* Treatment with another investigational drug within 4 weeks prior to enrollment
* History, or current suspicion of intussusception or ileus or gastrointestinal obstruction as per investigator's judgment
* Uncontrolled thyroid disease as per investigator judgment
* Hemoglobin or hematocrit < 75 percentage (%) of the lower limit of normal range
* Known severe or moderate hepatic impairment
* Clinical signs of hypotension that in the investigator's judgment would preclude initiation of a PAH-specific therapy
* Participants with severe renal insufficiency
* Known hypersensitivity to the investigational treatment or to any of the excipients of the drug formulations

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Boisson, Study Director — Actelion
Locations (34):
- United States (3):
  - Children'S Hospital Cardiac Care Center University Of Colorado, Aurora, Colorado
  - University of Iowa Hospital, Iowa City, Iowa
  - Seattle Children's Hospital, Seattle, Washington
- Belarus (2):
  - State Institution Republican Scientific And Practical Center For Pediatric Surgery, Minsk
  - Health Institution 4Th City Children'S Clinical Hospital, Minsk
- UZ Gent, Ghent, Belgium
- Centre Hospitalier Sainte Justine, Montreal, Quebec, Canada
- China (2):
  - Beijing Anzhen Hospital, Beijing
  - Shanghai Childrens Medical Center, Shanghai
- France (3):
  - CHU Arnaud de Villeneuve, Montpellier
  - Hôpital Necker - Enfants Malades, Paris
  - Chu Hopital Des Enfants, Toulouse
- Universitätsklinikum Freiburg Zentrum, Freiburg im Breisgau, Germany
- Gottsegen György Országos Kardiológiai Intézet, Felnőtt kardiológiai osztály, Budapest, Hungary
- Israel (2):
  - Schneider Children's Medical Center, Petach Tikvah
  - Sheba Medical Center, Ramat Gan
- Malaysia (2):
  - Sarawak Heart Center, Kota Samarahan
  - Institut Jantung Negara (National Heart Institute), Kuala Lumpur
- Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw, Poland
- Russia (6):
  - Kazan State Medical University, Kazan'
  - Federal State Budget Scientific Institution, Kemerovo
  - Moscow Scientific Research Institute For Pediatrics And Childrens Surgery Of Rosmedtechnologies, Moscow
  - Saint Petersburg State Pediatric Medical University, Saint Petersburg
  - Federal State Budgetary Institution, Saint Petersburg
  - Samara Regional Clinical Cardiological Dispensary, Samara
- Serbia (2):
  - Univerzitetska Dečja Klinika, Belgrade
  - Institut Za Zdravstvenu Zastitu Majke I Deteta Srbije Dr Vukan Cupic, Belgrade
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Ukraine (4):
  - Municipal Enterprise Of The Dnipropetrovsk Regional Council, Dnipro
  - State Institution Of The Ministry Of Health Of Ukraine, Kiev
  - Lviv Regional Clinical Hospital, Lviv
  - Municipal Institution Of The Zaporizhzhya Regional Council, Zaporizhzhya
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Beghetti M, Axelsen LN, Borissoff JI, Farhan M, Grill S, Leng S, Russu A, Lesage C, Remenova T, Hsu Schmitz SF, Moledina S. A prospective, multicenter, open-label, single-arm Phase 2 study to investigate the pharmacokinetics, safety, tolerability, and exploratory efficacy of selexipag in children with pulmonary arterial hypertension. Chest. 2025 Dec 20:S0012-3692(25)05947-1. doi: 10.1016/j.chest.2025.12.013. Online ahead of print. PMID 41429287

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years): Pediatric participants with pulmonary arterial hypertension (PAH) aged between >=12 to <18 years received Selexipag (Uptravi /ACT-293987/JNJ-67896049) orally on Day 1 based on body weight (>=50 kilograms [kg] with a starting dose of 200 micrograms [mcg] and up-titrated to individual maximum tolerated dose [iMTD] of up to 1,600 mcg; weight >=25 to <50 kg: with a starting dose of 150 mcg and up-titrated to the iMTD of up to 1200 mcg; weight >=9 to <25 kg at a starting dose of 100 mcg , up titrated to the iMTD of 800 mcg) twice daily during the first 12 weeks. Up-titration was followed by a stable maintenance treatment period from Week 12 up to end of treatment.
- Cohort 2 (>=6 to <12 Years): Pediatric participants with PAH aged between >=6 to <12 years received Selexipag (Uptravi /ACT-293987/JNJ-67896049) orally on Day 1 based on body weight (>=50 kilograms [kg] with a starting dose of 200 micrograms [mcg] and up-titrated to iMTD of up to 1,600 mcg; weight >=25 to <50 kg: with a starting dose of 150 mcg and up-titrated to the iMTD of up to 1200 mcg; weight >=9 to <25 kg at a starting dose of 100 mcg , up-titrated to the iMTD of up to 800 mcg) twice daily during the first 12 weeks. Up-titration was followed by a stable maintenance treatment period from Week 12 up to end of treatment.
- Cohort 3 (>=2 to <6 Years): Pediatric participants with PAH aged between >=2 to <6 years received Selexipag (Uptravi /ACT-293987/JNJ-67896049) orally on Day 1 based on body weight (>=50 kilograms [kg] with a starting dose of 200 micrograms [mcg] and up-titrated to iMTD of up to 1,600 mcg; weight >=25 to <50 kg: with a starting dose of 150 mcg and up-titrated to the iMTD of up to 1200 mcg; weight >=9 to <25 kg at a starting dose of 100 mcg , up-titrated to the iMTD of up to 800 mcg) twice daily during the first 12 weeks. Up-titration was followed by a stable maintenance treatment period from Week 12 up to end of treatment.
Period: Overall Study
Arm/Group | Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years) | Cohort 2 (>=6 to <12 Years) | Cohort 3 (>=2 to <6 Years)
Started | 22 | 21 | 20
Completed | 0 | 0 | 0
Not Completed | 22 | 21 | 20
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 3 | 0 | 3
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Other | 1 | 0 | 0
Not completed — Ongoing | 16 | 19 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years) | Cohort 2 (>=6 to <12 Years) | Cohort 3 (>=2 to <6 Years) | Total
Number analyzed (Participants) | 22 | 21 | 20 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.79) | 8.5 (1.36) | 3.8 (1.28) | 9 (4.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 10 | 36
  Male | 7 | 10 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 18 | 19 | 19 | 56
  Unknown or Not Reported | 3 | 2 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 6 | 7 | 16
  White | 16 | 12 | 11 | 39
  Unknown or Not Reported | 3 | 2 | 1 | 6
  Other | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  BELARUS | 4 | 2 | 3 | 9
  BELGIUM | 0 | 0 | 1 | 1
  CHINA | 0 | 1 | 7 | 8
  FRANCE | 3 | 1 | 1 | 5
  GERMANY | 0 | 1 | 0 | 1
  HUNGARY | 1 | 2 | 2 | 5
  ISRAEL | 0 | 1 | 2 | 3
  MALAYSIA | 3 | 4 | 0 | 7
  RUSSIAN FEDERATION | 7 | 0 | 2 | 9
  TAIWAN | 0 | 1 | 0 | 1
  UKRAINE | 1 | 4 | 0 | 5
  UNITED KINGDOM | 0 | 1 | 1 | 2
  UNITED STATES | 1 | 2 | 0 | 3
  Serbia | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve Over a Dose Interval at Steady State of Selexipag and Its Metabolite ACT-333679 Combined (AUCτ, ss, Combined)
Description: AUCτ, ss, combined was defined as the area under the plasma concentration-time curve over one dosing interval at steady state. AUCτ,ss,combined was calculated as 1/38 AUCτ,ss,selexipag plus 37/38 AUCτ,ss,ACT-333679.
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Population: The Pharmacokinetic analysis set included all participants from the safety set who complied with the protocol sufficiently and did not deviate from the protocol in a way that might affect the PK outcome of the study.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms*hour per milliliter
Arm/Group | Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years) | Cohort 2 (>=6 to <12 Years) | Cohort 3 (>=2 to <6 Years)
Number analyzed (Participants) | 21 | 21 | 17
nanograms*hour per milliliter | 21.56 [17.32 to 26.84] | 20.40 [16.83 to 24.73] | 18.57 [15.16 to 22.74]

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over a Dose Interval of Selexipag at Steady State (AUCτ,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Over a Dose Interval of ACT-333679 at Steady State (AUCτ,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Maximum Observed Plasma Concentration of Selexipag at Steady State (Cmax,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Maximum Observed Plasma Concentration of ACT-333679 at Steady State (Cmax,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration of Selexipag at Steady State (Tmax,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration of ACT-333679 at Steady State (Tmax,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Trough Concentration of Selexipag at Steady State (Ctrough,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Trough Concentration of ACT-333679 at Steady State (Ctrough,ss)
Time Frame: Week 1,Week 12: pre-dose, 1, 2, 4, 6, 8 and 12 h post-morning dose. Week 2, 4 and 6: pre-dose (Up to Week 12)
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (End of Treatment [EOT] + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs) (EOT + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Permanent Discontinuation of Study Drug
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Number of Participants With Treatment-emergent Deaths (EOT + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

14. Secondary Outcome: Number of Participants With Treatment-emergent Marked Laboratory Abnormalities (EOT + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

15. Secondary Outcome: Change From Baseline in Hematology Parameters (EOT + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

16. Secondary Outcome: Change From Baseline in Chemistry Parameters (EOT + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

17. Secondary Outcome: Number of Participants With Treatment-emergent Electrocardiogram (ECG) Abnormalities (EOT + 3 Days)
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

18. Secondary Outcome: Change From Baseline in Thyroid Stimulating Hormone (TSH) up to EOT + 3 Days
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

19. Secondary Outcome: Change From Baseline in Blood Pressure
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2027-12

20. Secondary Outcome: Change From Baseline in Heart Rate
Time Frame: Up to 7 years
Reporting Status: Not Posted, anticipated posting 2027-12

21. Secondary Outcome: Change From Baseline Over Time in Height up to EOT+3 Days
Time Frame: EOT+3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

22. Secondary Outcome: Change From Baseline Over Time in Body Mass Index (BMI) up to EOT + 3 Days
Time Frame: EOT+ 3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

23. Secondary Outcome: Change From Baseline in Sexual Maturation (Tanner Stage) up to End of Treatment (EOT + 3 Days)
Time Frame: EOT+ 3 days (Up to Week 17)
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: Up to 3 years 8 months
Description: The safety analysis set included all participants who received at least one dose of study treatment.
Arm/Group | Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years) | Cohort 2 (>=6 to <12 Years) | Cohort 3 (>=2 to <6 Years)
All-Cause Mortality (participants affected / at risk) | 3/22 | 0/21 | 3/20
Serious Adverse Events (participants affected / at risk) | 12/22 | 4/21 | 6/20
Other Adverse Events (participants affected / at risk) | 21/22 | 20/21 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years) (N=22) | Cohort 2 (>=6 to <12 Years) (N=21) | Cohort 3 (>=2 to <6 Years) (N=20)
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 2
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Covid-19 (Infections and infestations) | 4 | 1 | 0
Dengue Fever (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 1
Pneumonia Aspiration (Infections and infestations) | 0 | 0 | 1
Pneumonia Mycoplasmal (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Biopsy Kidney (Investigations) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brain Oedema (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2
Focal Segmental Glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Hypertensive Crisis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Suffocation Feeling (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wisdom Teeth Removal (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Greater Than or Equal to [>=] 12 Years to Less Than [<] 18 Years) (N=22) | Cohort 2 (>=6 to <12 Years) (N=21) | Cohort 3 (>=2 to <6 Years) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 1
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Anomalous Pulmonary Venous Connection (Congenital, familial and genetic disorders) | 1 | 0 | 0
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Delayed Puberty (Endocrine disorders) | 1 | 0 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 4 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 1 | 0
Gingival Swelling (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 6 | 2
Oesophageal Stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 9 | 7
Asthenia (General disorders) | 3 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 1
Chills (General disorders) | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 1
Exercise Tolerance Decreased (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 1
Influenza Like Illness (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 3 | 5 | 4
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 1 | 1
Blastocystis Infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 4 | 0 | 2
Dientamoeba Infection (Infections and infestations) | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Klebsiella Infection (Infections and infestations) | 0 | 0 | 1
Mycoplasma Infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 4 | 1 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Electric Shock (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Foreign Body in Ear (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Medication Error (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 1 | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0
N-Terminal Prohormone Brain Natriuretic Peptide Abnormal (Investigations) | 0 | 0 | 1
N-Terminal Prohormone Brain Natriuretic Peptide Increased (Investigations) | 2 | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0
Oxygen Saturation Decreased (Investigations) | 2 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 2
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 11 | 11 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Initial Insomnia (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Middle Insomnia (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Renal Cyst (Renal and urinary disorders) | 1 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea at Rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary Hypertensive Crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Androgenetic Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Medical Device Repositioning (Surgical and medical procedures) | 0 | 0 | 1
Ovarian Cystectomy (Surgical and medical procedures) | 1 | 0 | 0
Cyanosis (Vascular disorders) | 1 | 2 | 0
Flushing (Vascular disorders) | 5 | 2 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 1
Peripheral Coldness (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT03492177/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03492177/SAP_001.pdf